CLINICAL TRIAL: NCT01810536
Title: High Flow Nasal Oxygen for Children With Cystic Fibrosis Presenting With Respiratory Failure - a Randomized Controlled Study
Acronym: HIFLOWCF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It was impossible for us to include patients
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luiz Vicente Ribeiro Ferreira da Silva Filho, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIFLOWCF
Record Dates: First submitted 2013-03-08; First posted 2013-03-13 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; oxygen; respiratory failure
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hi-flow nasal cannula (Experimental): This group will receive supplemental oxygen by nasal cannula using the Optiflow system, with high flows of 100% humidified oxygen
  Interventions: Device: Hi-flow nasal cannula
- Venturi mask (Active Comparator): This group will receive supplemental oxygen by the current standard in our Institution: Venturi masks
  Interventions: Device: Venturi mask

INTERVENTIONS:
Device: Hi-flow nasal cannula — Different ways of providing supplemental oxygen will be compared: hi-flow nasal cannulas versus Venturi masks
  Other Names: Optiflow; MaxVenturi
  Arms: Hi-flow nasal cannula
Device: Venturi mask
  Arms: Venturi mask

SUMMARY:
Respiratory exacerbations are frequent among cystic fibrosis patients and supplemental oxygen is usually required. We will compare a new high flow nasal cannula system with Venturi masks for oxygen supplementation to patients with CF hospitalized for respiratory exacerbation.

DETAILED DESCRIPTION:
Introduction: Cystic fibrosis (CF) is a genetic disease that leads to chronic lung infections and recurrent respiratory exacerbations. Supplemental oxygen is usually required during respiratory exacerbations. Recently, a new high flow nasal cannula system that provides flows up to 40l/min at 100% humidification was developed and tested in neonates and children, providing greater comfort to the patient. The main hypothesis of the study is that this method has advantages for oxygen supplementation to patients with CF hospitalized for respiratory exacerbation. Methods: 40 patients with CF aged 6 to 18 years will be randomized to receive supplemental oxygen via nasal cannula or Venturi masks during hospitalization for respiratory exacerbation. Main outcomes will be the duration of hospitalization and oxygen supplementation, viscosity and transportability of sputum and personal impressions of patients regarding the method of oxygen administration (questionnaire). Spirometry and venous blood gas analysis will be performed after the second hospital day, and sputum samples will be obtained in the first and third day of hospitalization. Clinical treatment (antibiotics, etc) will be defined by the medical team of the institution, not involved in the study. Expected Results: The use of high flow nasal cannula will result in significantly less time of supplemental oxygen, with increased comfort for patients, without significant differences in the levels of PaCO2. Sputum samples obtained from the patients treated with the high flow nasal cannula will have lower viscosity and higher transportability as compared to those obtained from patients treated with Venturi mask.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of cystic fibrosis
* Age between 6 and 17 years
* Ability to perform lung function testing
* Hospital admission due to acute pulmonary exacerbation in the last 12h
* Regular use of Pulmozyme
* Need for high FiO2 defined as more than 2 liters per minute in the nasal cannula or need of a Venturi mask

Exclusion Criteria:

* Recent admission (less than 30 days)
* Recent or current atelectasis (less than 3 months)
* Hemoptysis or pneumothorax
* Need for a bronchoscopy during admission
* Need for non-invasive ventilation for more than 2 hours/day

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2013-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Oxygen supplementation period | up to 14 days
  Since most CF patients admitted due to a respiratory exacerbation need supplemental oxygen for up to 96h, we aim at a reduction of at least 12h in this period.

SECONDARY OUTCOMES:
Days in the hospital | Up to 14 days

OTHER OUTCOMES:
Time to recover the baseline forced expiratory volume in one second | Up to 14 days
  return to the baseline (stable) FEV1

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto da Criança, Hospital das Clínicas da FMUSP, São Paulo, Brazil